CLINICAL TRIAL: NCT01301157
Title: Study to Investigate the Efficacy and the Safety of M518101 in Plaque Psoriasis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maruho Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M518101-US01
Record Dates: First submitted 2011-02-18; First posted 2011-02-23 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-10

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — calcipotriene

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 25ug M518101 (Experimental)
  Interventions: Drug: M518101
- Vehicle (Placebo Comparator)
  Interventions: Drug: placebo
- Dovonex (Active Comparator)
  Interventions: Drug: Dovonex
- 50ug M518101 (Experimental)
  Interventions: Drug: M518101

INTERVENTIONS:
Drug: M518101 — Proper quantity twice a day
  Arms: 25ug M518101; 50ug M518101
Drug: placebo — Proper quantity twice a day
  Arms: Vehicle
Drug: Dovonex — Proper quantity twice a day
  Arms: Dovonex

SUMMARY:
This study is to evaluate the efficacy and safety of M518101 and the dose relationship among two doses of M518101 and placebo in male and female plaque psoriasis patients.

DETAILED DESCRIPTION:
This study is to evaluate the efficacy and safety of M518101 and the dose response relationship among two doses of M518101 and placebo in male and female plaque psoriasis patients and to confirm the persistence of the effect of M518101.

ELIGIBILITY:
Inclusion Criteria:

1. Who are able and willing to give signed informed consent
2. Who are male or females aged 18 years or older with plaque psoriasis confirmed by the Investigator.
3. Who have less than 20% of body surface area (BSA) afflicted with plaques
4. Who are neither pregnant nor breast-feeding, nor plan to become pregnant during the study.

Exclusion Criteria:

1. Who have a history of allergy to vitamin D3 derivative preparations.
2. Who have a history of relevant drug hypersensitivity.
3. Who have a history of contact dermatitis induced by a topical medicine.
4. Who are pregnant or lactating.
5. Who have any renal or hepatic insufficiency, or clinically significant cardiac, renal or hepatic disease.
6. Who are not deemed eligible as determined by medical history, physical examination or clinical laboratory safety tests.
7. Who have clinically relevant history or presence of any disease or surgical history other than psoriasis which is likely to affect the conduct of the study.
8. Whose serum calcium levels exceed the upper limit of reference range
9. Who have used any investigational medicinal product and/or participated in any clinical study within 60 days before the day of signing the ICF.
10. Who have been treated with systemic therapy within 2 weeks before the day of signing the ICF and during the wash-out period.
11. Who have been treated with biologics within 5 half-lives of the biologics before the day of randomization.
12. Who have been treated with topical therapy during the wash-out period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2011-02; Primary Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
severity of plaque psoriasis | 8 weeks after dosing

SECONDARY OUTCOMES:
Investigator global assessment | 8 weeks after dosing

CONTACTS AND LOCATIONS:
Locations (32):
- United States (32):
  - University of Alabama (UAB) Dermatology, Birmingham, Alabama
  - Coastal Carolina Research, Mobile, Alabama
  - Sierra Medical Research, Fresno, California
  - Therapeutics Clinical Research, San Diego, California
  - Clinical Science Institute, Santa Monica, California
  - Visions Clinical Research, Boynton Beach, Florida
  - Ameriderm Research, Jacsonville, Florida
  - Ameriderm Research, Ormond Beach, Florida
  - Atlanta Dermatology, Vein & Research Ctr, Alpharetta, Georgia
  - NorthShore University HealthSystem, Skokie, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - The Southbend Clinic, LLC, South Bend, Indiana
  - Derm Research, Louisville, Kentucky
  - Medical Development Centers, LLC, Baton Rouge, Louisiana
  - Medical Development Centers, LLC, Opelousas, Louisiana
  - Hamzavi Dermatology, Fort Gratiot, Michigan
  - Central Dermatology, St Louis, Missouri
  - Washington University, Dermatology Clinical Trials Unit, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Section of Dermatology, Lebanon, New Hampshire
  - Skin Search of Rochester, Inc., Rochester, New York
  - DermResearchCenter of New York, Inc, Stony Brook, New York
  - Dermatology Consulting Services, High Point, North Carolina
  - Wilmington Dermatology Center, Wilmington, North Carolina
  - Radiant Research, Columbus, Ohio
  - OUHSC-Dermatology, Oklahoma City, Oklahoma
  - Baker Allergy, Asthma and Dermatology Research Center, LLC, Lake Oswego, Oregon
  - Palmetto Clinical Trial Services, LLC, Greenville, South Carolina
  - Arlington Research Center, Inc, Arlington, Texas
  - Center for Clinical Studies, Texas Medical Center, Houston, Texas
  - Dermatology Clinical Research Center, San Antonio, Texas
  - Virginia Clinical Research Inc., Norfolk, Virginia
  - Dermatology Associates, Seattle, Washington